CLINICAL TRIAL: NCT05130970
Title: A Randomized, Double-blind, Placebo-controlled, Study to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics of Garadacimab in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Garadacimab Safety, Pharmacokinetics, and Pharmacodynamics in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL312_2002; 2021 003162 12 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-11-23 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Garadacimab (Experimental): Administered IV and SC
  Interventions: Drug: Garadacimab
- Placebo (Placebo Comparator): Administered IV and SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Garadacimab — Participants received garadacimab intravenous (IV) loading dose followed by 3 subcutaneous (SC) doses.
  Other Names: Factor XIIa antagonist monoclonal antibody; CSL312
  Arms: Garadacimab
Drug: Placebo — Participants received a matching placebo IV loading dose, followed by 3 SC doses.
  Arms: Placebo

SUMMARY:
This is a prospective, phase 2a, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to assess the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of garadacimab in subjects with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 40 years of age
* Documented diagnosis of IPF

Exclusion Criteria:

* History of clinically significant cardiovascular disease, including myocardial infarction, unstable ischemic heart disease, congestive heart failure, or angina during the 6 months before screening
* Sinoatrial or atrioventricular block, uncontrolled hypertension
* Active bleeding or current clinically significant coagulopathy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (47):
- United States (25):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates Clinical Trials AZ, Phoenix, Arizona
  - National Institute of Clinical Research, Huntington Beach, California
  - University of Southern California - Center for Advanced Lung Disease, Los Angeles, California
  - University of California Irvine, Orange, California
  - Meris Clinical Research, Brandon, Florida
  - Reliant Medical Research, Miami, Florida
  - US Associates in Research LLC, Miami, Florida
  - Lakes Research, Miami Lakes, Florida
  - Renstar Medical Research, Ocala, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Hannibal Clinic, Hannibal, Missouri
  - Weill Cornell Medical Center, New York, New York
  - Superior Clinical Research, Smithfield, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Temple University TMS, Philadelphia, Pennsylvania
  - Clinical Trial Center of Middle Tennesse, Franklin, Tennessee
  - Elite Medical Research, Dallas, Texas
  - Southwest Family Medicine Associates, Dallas, Texas
  - Baylor Scott and White Health - Advanced Lung Disease Specialists, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Royal Adelaide Hospital, Adelaide, Australia
- Austria (2):
  - Medizinische Univerität Graz, Graz
  - Kepler Universitätsklinikum, Linz
- Belgium (2):
  - Universitair Ziekenhuis (UZ) Leuven, Leuven
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
- Odense Universitetshospital - Lungemedicinsk Forskningsenhed, Odense, Denmark
- Germany (4):
  - Fachkrankenhaus Coswig GmbH, Coswig
  - Universitaetsklinikum Essen - Ruhrlandklinik (Westdeutsches Lungenzentrum), Essen
  - Medizinische Hochschule Hannover - Klinik für Pneumologie, Hanover
  - Petrus Krankenhaus Wuppertal, Wuppertal
- Azienda Ospedaliera Universitaria Ospedali Riuniti Foggia, Foggia, Italy
- Poland (3):
  - Centrum Medycyny Oddechowej Bialymstoku, Bialystok
  - Twoja Przychodnia Centrum Medyczne Nowa Sol, Nowa Sól
  - Centrum Badań Klinicznych NZOZ, Wroclaw
- Spain (2):
  - Giromed Institute, SLP, Barcelona
  - Hospital Universitario Puerta del Mar (HUPM), Cadiz
- United Kingdom (4):
  - The Churchill Hospital - Oxford University Hospitals NHS Trust, Oxford, MD
  - Queen Elizabeth Hospital, Birmingham
  - Altnagelvin Area Hospital, Londonderry
  - Manchester Univ NHS - Wythenshawe Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 47 study sites in 11 countries (Australia, Austria, Belgium, Canada, Denmark, Germany, Italy, Poland, Spain, the United Kingdom [UK], and the United States of America [USA]). No participants from Italy were enrolled in the study.
Pre-assignment Details: A total of 131 potential participants were screened for eligibility. Out of these, 81 participants met all selection criteria and were enrolled in the study, and 50 individuals failed to meet the selection criteria and were not enrolled in the study.
Period: Overall Study
Arm/Group | Garadacimab | Placebo
Started | 40 | 41
Completed | 38 | 36
Not Completed | 2 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Garadacimab: Participants received garadacimab IV loading dose followed by 3 SC doses.
- Total: Total of all reporting groups
Arm/Group | Garadacimab | Placebo | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.6 (6.19) | 72.9 (6.17) | 72.8 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 26 | 20 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 37 | 39 | 76
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 0 | 1
  Austria | 3 | 0 | 3
  Belgium | 0 | 3 | 3
  United States | 19 | 21 | 40
  Poland | 5 | 4 | 9
  Denmark | 3 | 2 | 5
  United Kingdom | 4 | 4 | 8
  Australia | 1 | 0 | 1
  Germany | 3 | 4 | 7
  Spain | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent (TE) Serious Adverse Events (SAEs)
Description: A TE SAE is defined as an SAE reported at or after the start of the first administration of study treatment. A SAE is defined as any untoward medical occurrence that at any dose results in: death, life-threatening event, initial or prolongation of existing hospitalization, disability or incapacity, congenital anomaly or birth defect, or any other medically significant event.
Time Frame: Up to 22 weeks
Population: This analysis was performed on the safety analysis set (SAS). The SAS was defined as all participants who received any portion of an IV infusion or SC injection of garadacimab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 5 | 2

2. Primary Outcome: Percentage of Participants With TE SAEs
Description: as for outcome 1
Time Frame: Up to 22 weeks
Population: This analysis was performed on the SAS. The SAS was defined as all participants who received any portion of an IV infusion or SC injection of garadacimab or placebo.
Measure: Number; unit: Percentage of participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Percentage of participants | 12.5 | 4.9

3. Primary Outcome: Number of Participants With TE Adverse Events of Special Interests (AESIs)
Description: The following TEAEs were considered as AESIs: Bleeding events that were abnormal in the opinion of the Investigator, Thromboembolic events (non-systemic thrombosis [e.g., localized thrombosis associated with vascular access] was not considered an AESI), and Severe hypersensitivity including anaphylaxis.
Time Frame: Up to 22 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 2 | 0

4. Primary Outcome: Percentage of Participants With TE-AESIs
Description: as for outcome 3
Time Frame: Up to 22 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Percentage of participants | 5.0 | 0

5. Primary Outcome: Number of Participants With Garadacimab Induced Anti Drug Antibodies (ADAs) in Plasma
Time Frame: At Day 36 and Day 92 after the first treatment
Population: This analysis was performed on the SAS. The SAS was defined as all participants who received any portion of an IV infusion or SC injection of garadacimab or placebo. Here, the Overall Number of Participants Analyzed (N) included all participants who were evaluated for this outcome measure and the Number Analyzed (n), included all participants who were evaluated for this outcome measure for the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 39 | 37
Participants
  At Day 36 | 1 | 2
  At Day 92: number analyzed (Participants) | 38 | 36
  At Day 92 | 1 | 1

6. Primary Outcome: Percentage of Participants With Garadacimab Induced ADAs in Plasma
Time Frame: At Day 36 and Day 92 after the first treatment
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 39 | 37
Percentage of participants
  At Day 36 | 2.6 | 5.4
  At Day 92: number analyzed (Participants) | 38 | 36
  At Day 92 | 2.6 | 2.8

7. Primary Outcome: Number of Participants With TE Clinically Significant Abnormalities in Laboratory Assessments Reported as Adverse Events (AEs)
Time Frame: Up to 14 weeks after treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 0 | 0

8. Primary Outcome: Percentage of Participants With TE Clinically Significant Abnormalities in Laboratory Assessments Reported as AEs
Time Frame: Up to 14 weeks after treatment
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 40 | 41
Percentage of participants | 0.0 | 0.0

9. Secondary Outcome: Trough Plasma Concentration (Ctrough) After SC Administration of Garadacimab
Time Frame: At Day 36 and Day 64
Population: This analysis was performed on pharmacokinetic analysis set (PKS). The PKS was defined as all participants in the SAS who received >= 1 dose of garadacimab with >= 1 measurable concentration of garadacimab after administration. Here, the Overall Number of Participants Analyzed (N) included all participants who were evaluated for this outcome measure and the Number Analyzed (n), included all participants who were evaluated for this outcome measure for the specified timepoint.
Measure: Mean (Standard Deviation); unit: Microgram/milliliter (ug/mL)
Arm/Group | Garadacimab
Number analyzed (Participants) | 37
Microgram/milliliter (ug/mL)
  At Day 36 | 16.445 (6.0362)
  At Day 64: number analyzed (Participants) | 35
  At Day 64 | 17.123 (7.9383)

10. Secondary Outcome: Maximum Plasma Concentration (Cmax) (Last SC Dosing Interval Only) of Garadacimab
Time Frame: After dosing on Day 64
Population: This analysis was performed on PKS. The PKS was defined as all participants in the SAS who received >= 1 dose of garadacimab with >= 1 measurable concentration of garadacimab after administration. Here, the Overall Number of Participants Analyzed (N) included all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Garadacimab
Number analyzed (Participants) | 38
ug/mL | 37.41 (15.507)

11. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) (Last SC Dosing Interval Only) of Garadacimab
Time Frame: After dosing on Day 64
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours (h)
Arm/Group | Garadacimab
Number analyzed (Participants) | 38
Hours (h) | 165.4585 [45.250 to 478.633]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Dose Interval (AUC0-tau) (Last SC Dosing Interval Only) of Garadacimab
Time Frame: After dosing on Day 64
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | Garadacimab
Number analyzed (Participants) | 29
h*ug/mL | 18094.6128 (6977.9036)

13. Secondary Outcome: Ctrough After IV Administration of Garadacimab
Time Frame: At Day 8
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Garadacimab
Number analyzed (Participants) | 36
ug/mL | 18.6054 (7.9685)

14. Secondary Outcome: Cmax After IV Administration of Garadacimab
Time Frame: After dosing on Day 1
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Garadacimab
Number analyzed (Participants) | 37
ug/mL | 79.636 (31.4406)

15. Secondary Outcome: Tmax After IV Administration of Garadacimab
Time Frame: After dosing on Day 1
Population: This analysis was performed on PKS. The PKS was defined as all participants in the SAS who received >= 1 dose of garadacimab with >= 1 measurable concentration of garadacimab after administration.
Measure: Median (Full Range); unit: h
Arm/Group | Garadacimab
Number analyzed (Participants) | 39
h | 0.1000 [0.017 to 0.967]

16. Secondary Outcome: Mean Change From Baseline in FXIIa-mediated Kallikrein Activity
Time Frame: Baseline and at Day 92
Population: This analysis was performed on pharmacodynamic analysis set (PDS). The PDS was defined as all participants in the SAS for whom analysis results were obtained for >= 1 of the exploratory biomarkers of interest. Here, the Overall Number of Participants Analyzed (N) included all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Nanomoles/liter/minutes (nmol/L/mins)
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 32 | 32
Nanomoles/liter/minutes (nmol/L/mins) | -0.0258 (0.0657) | 0.0072 (0.0706)

17. Secondary Outcome: Mean Percentage of Baseline in FXIIa-mediated Kallikrein Activity
Description: Percent baseline is calculated by using the formula visit value / baseline value multiplied by 100, percent baseline is reported as percentage in the outcome measure.
Time Frame: Baseline and at Day 92
Population: This analysis was performed on PDS. The PDS was defined as all participants in the SAS for whom analysis results were obtained for >= 1 of the exploratory biomarkers of interest. Here, the Overall Number of Participants Analyzed (N) included all participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent baseline
Arm/Group | Garadacimab | Placebo
Number analyzed (Participants) | 32 | 32
Percent baseline | 129.56 (215.689) | 124.83 (68.872)

ADVERSE EVENTS:
Time Frame: Up to 22 weeks
Description: This analysis was performed on SAS. The SAS was defined as all participants who received any portion of an IV infusion or SC injection of garadacimab or placebo.
Arm/Group | Garadacimab | Placebo
All-Cause Mortality (participants affected / at risk) | 1/40 | 1/41
Serious Adverse Events (participants affected / at risk) | 5/40 | 2/41
Other Adverse Events (participants affected / at risk) | 18/40 | 19/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Garadacimab (N=40) | Placebo (N=41)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Garadacimab (N=40) | Placebo (N=41)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (8)
Fatigue (General disorders) | 3 (4) | 3 (4)
Non-cardiac chest pain (General disorders) | 2 (3) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4) | 1 (1)
C-reactive protein increased (Investigations) | 1 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 4 (6)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (6)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT05130970/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT05130970/SAP_001.pdf